CLINICAL TRIAL: NCT04274660
Title: Evaluation of the Diabetes and WELLbeing (DWELL) Programme for People With Type 2 Diabetes
Brief Title: Evaluation of Diabetes and WELLbeing Programme
Acronym: DWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Medway Community Healthcare (Unknown); Blackthorn Trust (Unknown); Arteveldehogeschool (Unknown); Kinetic Analysis (Unknown); Centre Hospitalier de Douai (Other); The Health and Europe Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2S01-058 DWELL; 10065G00484 (Other: Canterbury Christ Church University)
Record Dates: First submitted 2020-02-05; First posted 2020-02-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Treated With Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Health

STUDY DESIGN:
Intervention Model Description: Participants will be invited to take part in the 12-week DWELL Programme (the intervention) based on their eligibility as per the inclusion criteria. They will all receive the psycho-social education element in addition to two motivational interviews. Each element will be evaluated alone and in combination.
  The non-intervention group will be recruited in one of two ways - they will either be people with type 2 diabetes who do not wish to participate in the 12-week programme, or they are receiving routine care (which, for UK participants, is a locally commissioned 6-week programme).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWELL Intervention (Experimental): People with type 2 diabetes participating in the 12-week DWELL (Diabetes and WELLbeing) Programme
  Interventions: Behavioral: DWELL (Diabetes and WELLbeing) Programme
- DWELL non-intervention/Control (No Intervention): People with type 2 diabetes who are receiving routine care from their GP and healthcare team. People with type 2 diabetes will continue to receive routine standard care. Routine care in this respect constitutes usual health and social care or any other nationally or locally commissioned education programmes

INTERVENTIONS:
Behavioral: DWELL (Diabetes and WELLbeing) Programme — 12-week psychoeducational programme
  Arms: DWELL Intervention

SUMMARY:
This study evaluates the impact of 'DWELL' - a 12-week psycho-social education programme designed to help people with type 2 diabetes to better self-manage their condition. Up to 600 patients will participate in the programme, while a non-intervention group will receive routine care for their diabetes

DETAILED DESCRIPTION:
The DWELL (Diabetes and WELLbeing) 12-week programme has been designed to incorporate specific elements of diabetes education and is underpinned by motivational interviewing to ensure it is tailored to individuals. Each of the four elements of the programme - education, nutrition, physical activity and wellbeing - have been carefully selected based on previous research into diabetes education. The Canterbury Christ Church University (CCCU) DWELL Team are responsible for the evaluation of DWELL, which will explore whether the combination of the programme elements is effective in improving self-management. Additionally, a process evaluation and cost effectiveness analysis will be conducted alongside participant outcomes

The programme will be delivered at five sites (two in the UK, one in Belgium, one in France, one in the Netherlands). The CCCU DWELL research team will be responsible for quality assurance, management and analysis of data, sample size assessment and reporting of adverse events. Each delivery site is responsible for adhering to their own Standard Operating Procedures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Over the age of 18

Exclusion Criteria:

* Under the age of 18
* Pregnant women
* Individuals who do not have the mental capacity to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in diabetes self-management as assessed by the Diabetes Self-Care Activities Measure | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in self-management and self-care will be measured using the Diabetes Self-Care Activities Measure at four time points. The SDSCA assesses aspects of the diabetes regimen. Higher scores indicate greater taking of prescribed medication and undertaking footcare regime.

SECONDARY OUTCOMES:
Change in quality of life as assessed by the Short Form Health Survey (SF-12) | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in health related quality of life will be measured using the Short Form Health Survey (SF-12) at four time points. SF-12 measures eight health domains to assess physical health (min 6, max 20 - higher scores indicate better physical health) and mental health (min 6, max 24 - higher scores indicate better mental health)
Change in levels of physical activity as assessed by the International Physical Activity Questionnaire (IPAQ) | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in levels of physical activity will be measured using the International Physical Activity Questionnaire (IPAQ) at four time points. IPAQ collects information on physical activity participation in three domains as well as sedentary behaviour. There is no min or max score - participants indicate how much exercise they do per week which is converted into MET minutes. Greater MET minutes indicate greater levels of physical activity.
Change in illness perception as assessed by the Illness Perception Questionnaire (IPQ-R) | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in perception and attitudes towards type 2 diabetes will be measured using the Illness Perception Questionnaire (IPQ-R) at four time points. IPQ-R measures an individual's beliefs and feelings about their illness. The IPQ-R is split into 7 sub-scales: Timeline (min 6, max 30 - higher scores indicate participants expect diabetes to last longer); Consequences (min 6, max 30 - higher scores indicate perceived worse consequences of diabetes); Personal Control (min 6, max 30 - higher scores indicate higher perceived control over diabetes); Treatment Control (min 5, max 25 - higher scores indicate higher perceived effect of treatment); Illness Coherence (min 5, max 25 - higher scores indicate better perceived understanding of illness); Timeline Cyclical (min 4, max 20 - higher scores indicate greater unpredictability of diabetes symptoms); Emotional Representations (min 6, max 30 - higher scores indicate more negative emotions associated with diabetes)
Change in psychosocial self-efficacy as assessed by the Diabetes Empowerment Scale (DES-SF) | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in self-efficacy will be measured using the Diabetes Empowerment Scale (DES-SF) at four time points. DES-SF measures changes in psychosocial self-efficacy. Minimum score is 8, max is 40. Higher scores indicate greater sense of empowerment to self-manage condition.
Change in eating behaviour as assessed by the Dutch Eating Behaviour Questionnaire (DEBQ) | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in eating behaviour will be measured using the Dutch Eating Behaviour Questionnaire (DEBQ) at four time points. DEBQ assesses three distinct eating behaviours in adults: Emotional Eating (min 10, max 50 - higher scores indicate the patient makes more effort to restrain eating) ; External Eating (min 13, max 65 - higher scores indicate patient eats more for emotional reasons); Restrained Eating (min 10, max 50 - higher scores indicate more motivated to eat by external factors, such as the smell and look of food)
Change in Body Mass Index (BMI) as assessed by height and weight | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in height and weight will be combined to report BMI in kg/m^2 where a lower score indicates an improvement for this outcome
Change in waist circumference | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in waist circumference will be measured and reported in cm where a lower measurement indicates an improvement for this outcome
Change in average blood glucose levels as assessed by Hemoglobin A1c levels (HbA1c) | Baseline, end of programme (3 months), 6 months after programme, 12 months after programme
  Changes in blood glucose (sugar) levels will be assessed by reports of HbA1c blood test results, where a lower score indicates improvement in this outcome
Quality Adjusted Life Years (QALYs) | 2.5 years
  Health related quality of life will be measured using the EuroQol Five Dimensions (EQ-5D-5L). The EQ-5D contains 5 sub-scales with a min score of 1 and max score of 3. Higher scores indicate worse mobility, worse ability to self-care, worse ability to perform usual activities, more pain and more anxiety. Utility values will also be multiplied by the time spent in each state to generate QALYs. 1 QALY is equivalent to perfect health while less than perfect health carries a QALY between 0 and 1. The higher the number of QALYs gained the better the health outcomes for people living with type 2 diabetes.
Cost effectiveness | 2.5 years
  The cost of Quality Adjusted Life Years (QALYs) of people with type 2 diabetes in the intervention group will be compared with the control group to illustrate cost effectiveness of the DWELL Programme

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Hatzidimitriadou, PhD, Principal Investigator — Canterbury Christ Church University
Locations (5):
- Arteveldehogeschool, Ghent, Belgium
- Centre Hosptalier Douai, Douai, France
- Kinetic Analysis, Breda, 's-Hertogenbosch, Netherlands
- United Kingdom (2):
  - Medway Community Healthcare, Gillingham, Kent
  - Blackthorn Trust, Maidstone, Kent

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participant data relating to results in publications with regards to primary and secondary outcome measures will be shared through publishing platforms. Anonymised individual participant datasets may be shared via a suitable public data repository. A final report of the evaluation study will be made available via the Canterbury Christ Church University DWELL Project web page.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It is anticipated that the study protocol will be published in a suitable academic journal by 31 December 2020. Individual participant data sets relating to the study will be made available via an appropriate data repository starting 6 months after formal publication of results.
  The final report of the evaluation study will be available on Canterbury Christ Church University DWELL Project web page by 31 March 2023.
Access Criteria: Anonymised participant data sets relating to publications will be shared through the control measures of the publishing journals, such as full access to subscribers.

REFERENCES:
- [Background] Hatzidimitriadou, E., Manship, S., Thompson, T., Morris, R., Moore, J. and Hulbert, S. 2023. Evalatuation study of the diabetes and welbeing (DWELL) - Report 1: Evaluation methodology. Canterbury, UK Canterbury Christ Church University.
- [Background] Hatzidimitriadou, E., Manship, S., Thompson, T., Morris, R., Moore, J., Hulbert, S. and Saloniki, E.-C. 2023. Evaluation study of diabetes and wellbeing (DWELL) - Report 2: Participant outcomes. Canterbury, UK Canterbury Christ Church University.
- [Background] Hatzidimitriadou, E., Manship, S., Thompson, T., Morris, R., Moore, J. and Hulbert, S. 2023. Evaluation study of Diabetes and Wellbeing (DWELL) - Report 3: Process evaluation. Canterbury Canterbury Christ Church University.
- [Background] Hatzidimitriadou, E., Manship, S., Thompson, T., Morris, R., Moore, J., Hulbert, S. and Saloniki, E.-C. 2023. Evaluation study of diabetes and wellbeing (DWELL) - Report 4: Workforce training and cost effectiveness. Canterbury. UK Canterbury Christ Church University.
- See also: Evaluation study of diabetes and wellbeing (DWELL) - Report 4: Workforce training and cost effectiveness — https://repository.canterbury.ac.uk/item/95w32/evaluation-study-of-diabetes-and-wellbeing-dwell-report-4-workforce-training-and-cost-effectiveness
- See also: Hatzidimitriadou, E., Manship, S., Thompson, T., Morris, R., Moore, J. and Hulbert, S. 2023. Evaluation study of Diabetes and Wellbeing (DWELL) - Report 3: Process evaluation. Canterbury Canterbury Christ Church University. — https://repository.canterbury.ac.uk/item/95w31/evaluation-study-of-diabetes-and-wellbeing-dwell-report-3-process-evaluation
- See also: Hatzidimitriadou, E., Manship, S., Thompson, T., Morris, R., Moore, J., Hulbert, S. and Saloniki, E.-C. 2023. Evaluation study of diabetes and wellbeing (DWELL) - Report 2: Participant outcomes. Canterbury, UK Canterbury Christ Church University. — https://repository.canterbury.ac.uk/item/95w2z/evaluation-study-of-diabetes-and-wellbeing-dwell-report-2-participant-outcomes
- See also: Evalatuation study of the diabetes and welbeing (DWELL) - Report 1: Evaluation methodology — https://repository.canterbury.ac.uk/item/95w2x/evalatuation-study-of-the-diabetes-and-welbeing-dwell-report-1-evaluation-methodology